CLINICAL TRIAL: NCT06987539
Title: A Phase 2 Open-label Multicenter Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Inebilizumab in Children From 2 Years to Less Than 18 Years of Age With Generalized Myasthenia Gravis (gMG)
Brief Title: A Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Inebilizumab in Children With Generalized Myasthenia Gravis (gMG)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240236; 2025-520993-20 (Other: EU CT Number)
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Generalized Myasthenia Gravis
Keywords: Generalized Myasthenia Gravis; Inebilizumab; AMG 335; Uplizna
MeSH Terms: conditions — Myasthenia Gravis | interventions — inebilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inebilizumab (Experimental): Inebilizumab will be administered intravenously (IV).
  Interventions: Drug: Inebilizumab

INTERVENTIONS:
Drug: Inebilizumab — Inebilizumab will be administered IV.

SUMMARY:
The primary objectives of this study are to characterize the pharmacokinetics (PK) and pharmacodynamics (PD) of inebilizumab administered in pediatric participants with gMG, and to assess the safety and tolerability of inebilizumab administered in pediatric participants with gMG.

ELIGIBILITY:
Inclusion Criteria

* Participant's legally authorized representative has provided informed consent when the participant is legally too young to provide informed consent and the participant has provided written assent based on local regulations and/or guidelines before any study-specific activities/procedures being initiated.
* Age ≥ 2 to < 18 years of age on the day of enrollment.
* Diagnosis of gMG defined as:

  * Positive serologic test for anti-acetylcholine receptor (AChR) or anti-muscle-specific tyrosine kinase (MuSK) antibody (Ab) titers as confirmed at screening (1 retest allowed), and
  * At least 1 of the following:

    * History of abnormal neuromuscular transmission test results demonstrated by single-fiber electromyography or repetitive nerve stimulation; or
    * History of positive anticholinesterase test (eg, edrophonium chloride test); or
    * Participant demonstrated improvement in gMG signs on oral cholinesterase inhibitors, as assessed by the treating physician; or
    * Clinical syndrome consistent with a diagnosis of gMG, and not otherwise explained by another condition.
* Myasthenia Gravis Foundation of America Clinical Classification Class II, III, or IV at the time of screening.
* Quantitative Myasthenia Gravis score of 11 or greater at screening.
* Participants may enter the study on:

  * Corticosteroids only, with no dose increase within 4 weeks prior to screening, or
  * One allowed non-steroidal immunosuppressive therapies (IST) (azathioprine, mycophenolate mofetil, or mycophenolic acid) with continuous use for at least 6 months prior to screening and no dose increase within 4 months prior to screening, or
  * Combination of (1) corticosteroids with no dose increase within 4 weeks prior to screening and (2) one allowed non-steroidal IST with continuous use for at least 6 months prior to screening and no dose increase within 4 months prior to screening.
* Participants may enter the study on a stable dose of acetylcholinesterase inhibitors (pyridostigmine dose). The acetylcholinesterase inhibitor dose must have been stable for at least 2 weeks prior to enrollment.
* Vital signs and laboratory parameters within the normal ranges at screening, or, if outside normal ranges, deemed not clinically significant by the investigator.

Exclusion Criteria

* Thymectomy within 12 months prior to baseline (Day 1) visit or planned thymectomy during the duration of the treatment period.
* Unresected thymoma- Participants with benign thymoma resected > 12 months prior to screening may enroll.
* History of recurrent significant infections.
* Known immunodeficiency disorder, including current infection or positive test for human immunodeficiency virus (HIV).
* Positive test for chronic hepatitis B infection at screening.
* History of untreated hepatitis C infection, or positive antibody test for hepatitis C virus (HCV).
* History of active or latent tuberculosis (TB), or a positive QuantiFERON®-TB Gold test at screening, unless treatment for TB was completed per local guidelines.
* Receipt of any biologic B-cell-depleting therapy (eg, rituximab, ocrelizumab, obinutuzumab, ofatumumab, inebilizumab) or any experimental B-cell-depleting agent in the 6 months prior to screening.
* Receipt of any other monoclonal antibody (mAb) or large molecule biologic, including but not limited to FcRn inhibitors, anti-TNF mAbs, anti-janus kinase (JAK) Stat mAbs, and complement inhibitors within 6 months prior to screening.
* Participants who are pregnant or breastfeeding or planning to get pregnant.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2030-03-13 (Estimated); Study Completion 2030-03-13 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Inebilizumab | Up to Week 52
Area Under the Concentration-time Curve (AUC) of Inebilizumab | Up to Week 52
Half-life (t1/2) of Inebilizumab | Up to Week 52
Clearance (CL) of Inebilizumab | Up to Week 52
Volume of Distribution at Steady State (Vss) of Inebilizumab | Up to Week 52
Change from Baseline in Cluster of Differentiation 20 (CD20)+ B-cell Counts | Baseline and Week 78
Number of Participants Experiencing Treatment-emergent Adverse Events | Up to Week 78
Number of Participants Experiencing Clinically Significant Changes in Laboratory Parameters | Up to Week 78
Number of Participants Experiencing Clinically Significant Changes in Vital Signs | Up to Week 78

SECONDARY OUTCOMES:
Change from Baseline in Quantitative Myasthenia Gravis (QMG) Score | Baseline and Week 78
Change from Baseline in Myasthenia Gravis Activities of Daily Living (MG-ADL) Score | Baseline and Week 78
Change from Baseline in Euro Quality of Life-5 Dimension Youth (EQ-5D-Y) Score | Baseline and Week 78
Change from Baseline in Neurological Quality of Life (Neuro-QoL) Paediatric Fatigue Score | Baseline and Week 78
Number of Participants with Anti-drug Antibodies (ADAs) Present | Up to Week 78

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Austin Neuromuscular Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com